CLINICAL TRIAL: NCT00331539
Title: Relationship Between Auto NRT and Behavioural T & C Levels With the Nucleus Freedom Cochlear Implant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BnaiZionMC-06-ML-002-CTIL
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2005-07

CONDITIONS: Hearing Loss
Keywords: Cochlear implant; threshold (T) measurement; comfort (C) level; profound hearing loss; auditory stimuli; profound hearing loss patients eligible for the study should be capable of providing reliable; subjective counted thresholds and has good NRT recordings, implanted with; the Nucleus Freedom system
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

INTERVENTIONS:
Device: Cochlear Implant

SUMMARY:
Cochlear implants require programming on an individual basis to provide appropriate levels of electrical stimulation. This program, or "map", is placed in the speech processor of the cochlear implant. Success of implantation largely depends on the adequacy of this map. Cochlear implant fitting remains a difficult challenge in congenitally or pre-linguistically deafened children. It requires competence of experienced audiologists with expertise in behavioral techniques for hearing function assessment.Our goal is to establish the offset correlation between objective measurements (NRT and ESRT) and the behavioral measurements of T & Cs in different stimulation rates in the Freedom SP System.

DETAILED DESCRIPTION:
An open trail. The implantees will go through their routine programming sessions after implantation, the specified data will be collected and analyzed in order to establish the offset correlation which we seek for.

ELIGIBILITY:
Inclusion Criteria:Patients eligible for the study should be capable of providing reliable subjective counted thresholds (e.g. children older than 12 years of age at CI or adults) and has good NRT recordings, implanted with the Nucleus Freedom system

-

Exclusion Criteria:Implantees With any other serious illness, Who can not give a reliable subjective counted thresholds

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2008-06

PRIMARY OUTCOMES:
To find possible correlation between behavioral counted T & C levels at different stimulation rates and NRT thresholds using the Auto NRT and ESRT over time, from switch on up to 12 months period.
To find possible changes over time in NRT thresholds (12 months period).
To find possible changes over time in ESRT thresholds (9 months period) starting 3 months post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Luntz, MD, Principal Investigator — Head of the E.N.T department head and neck surgery Bnai Zion MC ISRAEL
Locations (1):
- Bnai Zion MC, Haifa, Israel